CLINICAL TRIAL: NCT03085732
Title: The Effect of Intraabdominal Saline Irrigation on Infectious Morbidities and Gastrointestinal Outcomes in Patients Undergoing Abdominal Hysterectomies for Benign Causes
Brief Title: The Effect of Intraabdominal Saline Irrigation in Abdominal Hysterectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadiye Koroglu, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nadiye Koroglu
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Gynecologic Surgery
Keywords: saline irrigation; abdominal hysterectomy; postoperative infectious morbidities; gastrointestinal disturbances
MeSH Terms: interventions — Therapeutic Irrigation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation with saline solution (Active Comparator): during abdominal hysterectomy after vaginal cuff closure abdominal saline irrigation will be done
  Interventions: Drug: Irrigation with Saline Solution
- control (No Intervention): routine abdominal hysterectomy will be performed and no abdominal saline irrigation

INTERVENTIONS:
Drug: Irrigation with Saline Solution — During hysterectomy after vaginal cuff closure 500-1000 mL saline irrigation will be done.
  Arms: Irrigation with saline solution

SUMMARY:
The objective of this prospective randomised clinic study is to investigate the effect of peritoneal cavity saline irrigation during abdominal hysterectomies on postoperative infectious morbidities and gastrointestinal disturbance. The participants will be randomised to either an irrigation of abdominal cavity or the control group after vaginal closure. Assignment to one of the two treatment groups will be determined using a computer generated random numbers. Primary outcome is the rate of postoperative infectious morbidities. Secondary outcome is the rate of gastrointestinal disturbances (nausea, vomiting), use of antiemetic drugs and pain score in the postoperative period. 100 patients in each treatment arm planned.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hysterectomies for benign causes

Exclusion Criteria:

* patients who have diabetes mellitus patients undergoing hysterectomy for pelvic inflammatory disease or tuboovarian abscess

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-31 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative infectious morbidities | 10 day after hysterectomy operation
  vaginal cuff infection diagnosed with vagen cuff culture

SECONDARY OUTCOMES:
gastrointestinal outcomes: nausea by questionnaire | postoperative first day
  nausea by questionnaire
gastrointestinal outcome: vomiting by questionnaire | postoperative first day
  vomiting by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No